CLINICAL TRIAL: NCT03818880
Title: A Sub-Study to Assess the Choroidal Response to Novel Spectacle Lens to Control Myopia Progression (CHERRY)
Brief Title: Choroidal Response to Novel Spectacle Lens to Control Myopia Progression
Acronym: CHERRY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/654/18/SG
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myopia, Progressive
Keywords: Myopia; Myopia control
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Subjects wearing novel spectacle lenses will be assessed
  Interventions: Device: Novel spectacle lens design

INTERVENTIONS:
Device: Novel spectacle lens design — Spectacle lens to control progression of myopia

SUMMARY:
Diurnal variations in the thickness of the choroid have been reported in the literature, and, more recently, the role of the choroid has been studied with respect to its role in myopia (near-sightedness) progression.

DETAILED DESCRIPTION:
Diurnal variations in the thickness of the choroid have been reported in the literature , and, more recently, the role of the choroid has been studied with respect to its role in myopia (near-sightedness) progression. SightGlass Vision, Inc is conducting a multi-site, randomized, controlled, interventional study to confirm the efficacy and safety of spectacle lenses designed to inhibit the progression of myopia by reducing image contrast in peripheral vision. CORE is participating as a clinical site in this three year study which aims to compare changes in ocular length and cycloplegic auto-refraction in children randomised to wear one of either two test or one control spectacle lens designs; the CPRO-1802-001 (Cypress_SG) study. The sponsor is interested in conducting choroidal thickness measurements only at CORE's site by inviting those participants who have already been found eligible for the CPRO-1802-001 study to participate in this parallel study.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the CPRO-1802-001 (Cypress_SG) study at CORE
* Read and signed an Assent and their parent/guardian has signed an information consent letter

Exclusion Criteria:

* Transient health condition which may affect the eye(s) (e.g. a common cold, active allergies, fatigue, etc;)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 3 years
  Measurement of choroidal thickness by Triton optical coherence tomographer (OCT), including post-imaging analysis

SECONDARY OUTCOMES:
Visual field | 3 years
  Assessment of visual field to determine if changes in peripheral visual function by Humphrey Visual Field Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education, Canada; Jill Woods, BSc, MCOptom, Study Director — Centre for Ocular Research & Education, Canada
Locations (1):
- Centre for Ocular Research and Education, Waterloo, Ontario, Canada